CLINICAL TRIAL: NCT03601897
Title: An Open-Label, Multicenter, Phase 1b/2 Study of Rebastinib (DCC-2036) in Combination With Paclitaxel to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1b/2 Study of Rebastinib (DCC-2036) in Combination With Paclitaxel in Patients With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development program terminated.
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2036-01-003
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumor
Keywords: rebastinib; paclitaxel; breast cancer; ovarian cancer; endometrial cancer; gynecological carcinosarcoma; malignant mixed Mullerian tumor (MMMT)
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Carcinosarcoma | interventions — rebastinib; DCC-2036; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose escalation of rebastinib 50 milligram (mg) twice daily (BID) orally (PO) in combination with paclitaxel administered by intravenous (IV) infusion at 80 mg/meter squared (m^2) on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose escalation of rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in triple-negative breast cancer (TNBC). Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in TNBC. Rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in inflammatory breast cancer. Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in inflammatory breast cancer. Rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in ovarian cancer. Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in ovarian cancer. Rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in endometrial cancer. Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in endometrial cancer. Rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (Experimental): Dose expansion in gynecological carcinosarcoma (GCS). Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Rebastinib — Administered orally
  Other Names: DCC-2036
Drug: Paclitaxel — Paclitaxel administered by IV infusion at 80 mg/m^2

SUMMARY:
This is an open-label Phase 1b/2 multicenter study of rebastinib (DCC-2036) in combination with paclitaxel designed to evaluate the safety, tolerability, and pharmacokinetics (PK) in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age at the time of informed consent
2. Part 1 Histologically confirmed diagnosis of a locally advanced or metastatic solid tumor for which paclitaxel is considered appropriate treatment
3. Part 2

   * Triple-negative and Stage IV inflammatory breast cancer
   * Recurrent ovarian cancer
   * Recurrent, metastatic or high-risk endometrial cancer
   * Advanced (stage III or IV), or recurrent gynecological carcinosarcoma

     * Homologous or heterologous type carcinosarcoma (malignant mixed Mullerian tumor [MMMT] allowed
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of ≤2
5. Able to provide an archival tumor tissue sample
6. Adequate organ function and bone marrow reserve
7. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment
8. Patient must provide signed consent to participate in the study and is willing to comply with study-specific procedures

Exclusion Criteria:

1. Received prior anticancer or other investigational therapy within 28 days or 5× the half-life prior to the first dose
2. Not recovered from prior-treatment toxicities to Grade ≤1
3. Peripheral neuropathy of any etiology >Grade 1
4. Concurrent malignancy
5. Known active central nervous system (CNS) metastases
6. Use of systemic corticosteroids
7. Known retinal neovascularization, macular edema or macular degeneration
8. History or presence of clinically relevant cardiovascular abnormalities
9. QT interval corrected by Fridericia's formula (QTcF) >450 ms in males or >470 ms in females
10. Left ventricular ejection fraction (LVEF) <50% at screening
11. Arterial thrombotic or embolic events
12. Venous thrombotic event
13. Active infection ≥Grade 3
14. Human immunodeficiency virus (HIV) or hepatitis C (HCV) infection only if taking medications excluded per protocol, active hepatitis B (HBV), or active HCV infection
15. Use of proton pump inhibitors
16. If female, the patient is pregnant or lactating
17. Major surgery 4 weeks prior to the first dose of study drug
18. Malabsorption syndrome or other illness which could affect oral absorption
19. Known allergy or hypersensitivity to any component of rebastinib or any of its excipients.
20. Any other clinically significant comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Colorado Denver- Anschutz Medical Center, Aurora, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The University of Kansas Clinical Research Center, Kansas City, Kansas
  - Dana-Farber, Boston, Massachusetts
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants- Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Started | 24 | 19 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20
mITT Population (Modified Intent-to-Treat (mITT) Population includes all participants who had at least one dose of the combined study drugs, had measurable disease at baseline, and had at least one post-baseline assessment. Participants without a post-baseline assessment who discontinued study treatment due to clinical progression, death, or a rebastinib-related AE will also be included in the mITT population.) | 18 | 14 | 10 | 6 | 13 | 4 | 26 | 9 | 20 | 14 | 19
Completed | 1 | 6 | 5 | 4 | 9 | 2 | 12 | 5 | 9 | 5 | 7
Not Completed | 23 | 13 | 7 | 2 | 6 | 3 | 16 | 5 | 13 | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2: Dose escalation of rebastinib 50 mg BID PO in combination with paclitaxel administered by IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
- Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2: Dose expansion in TNBC. Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
- Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2: Dose expansion in ovarian cancer. Rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 24 | 19 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 14 | 7 | 4 | 14 | 4 | 15 | 8 | 7 | 9 | 6 | 106
  >=65 years | 6 | 5 | 5 | 2 | 1 | 1 | 13 | 2 | 15 | 7 | 14 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20 | 168
  Male | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 1 | 1 | 2 | 0 | 4 | 0 | 3 | 2 | 6 | 26
  White | 19 | 15 | 11 | 4 | 11 | 5 | 20 | 9 | 16 | 13 | 13 | 136
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 24 | 19 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20 | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants (pts) who experienced serious adverse events (SAE) and adverse events (AE).
Time Frame: Baseline up to 2.89 years
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 24 | 19 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20
Participants
  Any SAE | 16 | 12 | 3 | 3 | 2 | 3 | 9 | 5 | 10 | 9 | 9
  Any AE | 24 | 18 | 12 | 6 | 15 | 5 | 28 | 10 | 22 | 16 | 20

2. Primary Outcome: Objective Response Rate (ORR) (Part 2 Expansion)
Description: Percentage of participants who achieved an objective response of Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumor (RECIST) v1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline, or the appearance of one or more new lesions.
Time Frame: Baseline to PD or Death due to Any Cause (Up to 1.54 years)
Population: Part 2 mITT participants that were evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 10 | 6 | 13 | 4 | 26 | 9 | 20 | 14 | 19
percentage of participants | 0 [0.0 to 25.9] | 16.7 [0.9 to 58.2] | 7.7 [0.4 to 31.6] | 25.0 [1.3 to 75.1] | 30.8 [16.3 to 48.7] | 11.1 [0.6 to 42.9] | 20.0 [7.1 to 40.1] | 35.7 [15.3 to 61.0] | 5.3 [0.3 to 22.6]

3. Secondary Outcome: Objective Response Rate (ORR) (Part 1 Escalation)
Description: Percentage of pts who achieved an objective response of Complete Response (CR) or Partial Response (PR). Per RECIST v1.1, CR defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to have reduction in short axis to <10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or the appearance of one or more new lesions. Modified RECIST (mRECIST) used for pleural mesothelioma defines CR as the disappearance of any intratumoural arterial enhancement in all target lesions; PR as at least a 30% decrease in the sum of diameters of viable target lesions, taking as reference the baseline sum of the diameters of target lesions; PD as an increase of at least 20% in the sum of the diameters of viable target les
Time Frame: Baseline to PD or Death due to Any Cause (Up to 0.92 years)
Population: Part 1 mITT participants that were evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 18 | 14
percentage of participants | 16.7 [4.7 to 37.7] | 21.4 [6.1 to 46.6]

4. Secondary Outcome: Duration of Response (DOR)
Description: Time from CR or PR to the earliest documented evidence of PD or death due to any cause. Per RECIST v1.1, CR defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to have reduction in short axis to <10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or the appearance of one or more new lesions. mRECIST used for pleural mesothelioma defines CR as the disappearance of any intratumoural arterial enhancement in all target lesions; PR as at least a 30% decrease in the sum of diameters of viable target lesions, taking as reference the baseline sum of the diameters of target lesions; PD as an increase of at least 20% in the sum of the diameters of viable target lesions.
Time Frame: Time from CR or PR to PD or Death due to Any Cause (Up to 1.54 years)
Population: mITT participants that had CR or PR and were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 3 | 3 | 0 | 1 | 1 | 1 | 8 | 1 | 4 | 5 | 1
months | 11.1 [NA to NA] — The 90% Confidence Interval (CI) was not estimable due to insufficient number of events. | NA [NA to NA] — DOR median and 90% CI were not estimable due to insufficient number of events. |  | 6.9 [NA to NA] — The 90% CI was not estimable due to insufficient number of events. | 7.4 [NA to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [NA to NA] — DOR median and 90% CI were not estimable due to insufficient number of events. | 6.5 [5.4 to NA] — The 90% CI was not estimable due to insufficient number of events. | 5.5 [NA to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [4.6 to NA] — DOR median and 90% CI were not estimable due to insufficient number of events. | 8.8 [7.4 to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [NA to NA] — DOR median and 90% CI were not estimable due to insufficient number of events.

5. Secondary Outcome: Time to Progression (TTP)
Description: Time from first dose of study drug to the earliest documented evidence of PD. Per RECIST v1.1, PD defined as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions. mRECIST used for pleural mesothelioma defines PD as an increase of at least 20% in the sum of the diameters of viable target lesions.
Time Frame: First Dose of Study Drug to PD (Up to 2.61 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 18 | 14 | 10 | 6 | 13 | 4 | 26 | 9 | 20 | 14 | 19
months | 14.7 [3.7 to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [1.8 to NA] — TTP median and 90% CI were not estimable due to insufficient number of events. | 6.4 [1.8 to NA] — The 90% CI was not estimable due to insufficient number of events. | 5.3 [1.3 to 8.7] | 3.7 [1.9 to 6.4] | NA [1.8 to NA] — TTP median and 90% CI were not estimable due to insufficient number of events. | 9.1 [7.2 to 17.3] | 9.0 [3.6 to NA] — The 90% CI was not estimable due to insufficient number of events. | 6.2 [3.7 to NA] — The 90% CI was not estimable due to insufficient number of events. | 9.4 [5.5 to 12.0] | 3.5 [1.8 to 3.8]

6. Secondary Outcome: Progression-free-survival (PFS)
Description: Time from first dose of study drug to the earliest documented evidence of PD or death due to any cause. Participants who undergo surgical resection of target or non-target lesions, who have received other anticancer treatments, including surgical resection or radiation (other than palliative radiation to pre-existing bone metastases'), or who do not have a documented date of progression or death due to any cause will be censored at the date of the last assessment. PD per RECIST v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions. mRECIST used for pleural mesothelioma defines PD as an increase of at least 20% in the sum of the diameters of viable target lesions.
Time Frame: First Dose of Study Drug to PD or Death due to Any Cause (Up to 2.61 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2: Dose expansion in triple-negative breast cancer (TNBC). Rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 18 | 14 | 10 | 6 | 13 | 4 | 26 | 9 | 20 | 14 | 19
months | 6.5 [3.7 to 14.7] | NA [1.7 to NA] — PFS median and 90% CI were not estimable due to insufficient number of events. | 6.4 [1.8 to NA] — The 90% CI was not estimable due to insufficient number of events. | 5.3 [1.3 to 8.7] | 3.7 [1.9 to 6.4] | NA [1.8 to NA] — PFS median and 90% CI were not estimable due to insufficient number of events. | 9.1 [7.2 to 17.3] | 7.7 [3.6 to NA] — The 90% CI was not estimable due to insufficient number of events. | 6.2 [1.8 to NA] — The 90% CI was not estimable due to insufficient number of events. | 9.4 [5.5 to 12.0] | 3.5 [1.8 to 3.8]

7. Secondary Outcome: Overall Survival (OS)
Description: Time from first dose of study drug to date of death due to any cause. Participants who were still alive or who were lost to follow-up will be censored at the date of last contact.
Time Frame: First Dose of Study Drug to Death due to Any Cause (Up to 2.82 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 18 | 14 | 10 | 6 | 13 | 4 | 26 | 9 | 20 | 14 | 19
months | NA [5.2 to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [5.4 to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [6.3 to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [5.1 to NA] — OS median and 90% CI were not estimable due to insufficient number of events.

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Rebastinib (Part 1)
Description: Measure the Cmax
Time Frame: Part 1: Cycle 1 Day 1 (C1 D1), C1 D15 (Cycle = 28 days)
Population: Part 1 participants who received any study drug and had evaluable Cmax data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 24 | 19
nanograms/milliliter (ng/mL)
  Cycle 1 Day 1 | 77.4 (67.7) | 132 (76.4)
  Cycle 1 Day 15: number analyzed (Participants) | 19 | 15
  Cycle 1 Day 15 | 89.7 (80.1) | 143 (47.6)

9. Secondary Outcome: PK: Area Under the Concentration-time Curve (AUC) 0-6 Hours of Rebastinib (Part 1)
Description: Measure the AUC 0-6 hours
Time Frame: Part 1: Cycle 1 Day 1 (C1 D1), C1 D15 (Cycle = 28 days)
Population: Part 1 participants who received any study drug and had evaluable AUC data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanograms per hour (h*ng/mL)
Groups:
- Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2: Dose escalation of rebastinib 50 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
- Part 1 Arm 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2: Dose escalation of rebastinib 100 mg BID PO in combination with paclitaxel IV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 24 | 19
Hour times nanograms per hour (h*ng/mL)
  Cycle 1 Day 1 | 204 (67.9) | 337 (83.9)
  Cycle 1 Day 15: number analyzed (Participants) | 18 | 15
  Cycle 1 Day 15 | 283 (80.8) | 457 (56.6)

ADVERSE EVENTS:
Time Frame: Baseline up to 2.89 years
Groups:
- Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2: Dose expansion in inflammatory breast cancer. Rebastinib 50 mg BID PO in combination with paclitaxelIV infusion at 80 mg/m^2 on days 1, 8, and 15 of repeated 28-day cycles.
Arm/Group | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 7/24 | 4/19 | 0/12 | 1/6 | 1/15 | 0/5 | 0/28 | 2/10 | 2/22 | 0/16 | 3/20
Serious Adverse Events (participants affected / at risk) | 16/24 | 12/19 | 3/12 | 3/6 | 2/15 | 3/5 | 9/28 | 5/10 | 10/22 | 9/16 | 9/20
Other Adverse Events (participants affected / at risk) | 23/24 | 15/19 | 12/12 | 6/6 | 15/15 | 5/5 | 28/28 | 10/10 | 22/22 | 16/16 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=24) | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=19) | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=12) | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=6) | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=15) | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=5) | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=28) | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=10) | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=22) | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=16) | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=20)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=24) | Part 1 Arm 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=19) | Part 2 Cohort 1 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=12) | Part 2 Cohort 1 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=6) | Part 2 Cohort 2 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=15) | Part 2 Cohort 2 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=5) | Part 2 Cohort 3 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=28) | Part 2 Cohort 3 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=10) | Part 2 Cohort 4 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=22) | Part 2 Cohort 4 Rebastinib 100 mg + Paclitaxel 80 mg/m^2 (N=16) | Part 2 Cohort 5 Rebastinib 50 mg + Paclitaxel 80 mg/m^2 (N=20)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 5 (11) | 1 (3) | 3 (3) | 2 (2) | 2 (3) | 5 (13) | 2 (9) | 1 (1) | 5 (6) | 8 (28)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid cyst (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 4 (7) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (5) | 3 (3) | 2 (2)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 3 (4) | 1 (2) | 5 (5)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 10 (15) | 2 (3) | 3 (3) | 1 (1) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (16) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (6) | 2 (2) | 2 (2) | 5 (12) | 1 (2) | 11 (15) | 1 (2) | 7 (10) | 9 (13) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (8) | 1 (1) | 2 (3) | 7 (9) | 2 (2) | 6 (10) | 6 (6) | 5 (12) | 5 (8) | 8 (13)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 10 (11) | 4 (4) | 4 (4) | 5 (5) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (8) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 3 (3) | 2 (3) | 3 (3) | 7 (12) | 1 (1) | 11 (17) | 4 (4) | 11 (12) | 3 (9) | 8 (8)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (8) | 4 (4) | 3 (3) | 3 (5) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 5 (7) | 3 (4) | 1 (1) | 6 (14) | 6 (6)
Asthenia (General disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (12) | 6 (10) | 7 (9) | 4 (7) | 9 (10) | 2 (4) | 17 (21) | 5 (9) | 12 (21) | 7 (10) | 7 (13)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 13 (27) | 4 (7) | 10 (13) | 7 (12) | 7 (8)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (6) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 4 (8) | 4 (4) | 2 (3) | 2 (2) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (10) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site rash (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (3)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Intraocular pressure increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 6 (6) | 2 (3) | 5 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 1 (4) | 1 (1) | 1 (1) | 4 (9)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (10) | 0 (0) | 2 (2) | 1 (4) | 2 (7)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (4)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 3 (3) | 4 (5) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 4 (4) | 3 (5) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 5 (12) | 3 (4) | 6 (8) | 5 (6) | 3 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 8 (12) | 1 (2) | 4 (7) | 6 (9) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 1 (1) | 7 (7) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 6 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0) | 0 (0) | 2 (6) | 2 (2) | 3 (4) | 7 (10) | 4 (5) | 2 (2) | 6 (10) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (5) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 6 (7) | 3 (3) | 2 (5) | 2 (4) | 0 (0) | 13 (25) | 2 (2) | 11 (18) | 4 (5) | 4 (10)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (5) | 1 (2) | 4 (4) | 2 (3) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 5 (6) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 5 (8) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 7 (10) | 2 (2) | 9 (12) | 3 (4) | 3 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Paranasal sinus hyposecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6) | 2 (2) | 2 (3) | 5 (5) | 2 (3) | 14 (18) | 2 (2) | 5 (5) | 6 (7) | 6 (7)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 10 (20) | 3 (3) | 3 (3) | 4 (7) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial terminated on May 23, 2022, due to development program termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT03601897/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03601897/SAP_001.pdf